CLINICAL TRIAL: NCT00108797
Title: NovoSeven® (rFVIIa) by Single Dose for Home Treatment of Joint Bleeds in Haemophilia Patients With Inhibitors: A Pilot, Double-Blind Study Versus Standard Multiple Doses of NovoSeven® and Open-Label FEIBA®
Brief Title: Trial of NovoSeven® in Haemophilia - Joint Bleeds
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: F7HAEM-2068
Record Dates: First submitted 2005-04-18; First posted 2005-04-19 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A With Inhibitors; Haemophilia B With Inhibitors
MeSH Terms: interventions — Factor VII; anti-inhibitor coagulant complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: eptacog alfa (activated)
  Other Names: activated recombinant human factor VII
Drug: Feiba VH

SUMMARY:
This trial is conducted in the United States of America (USA). This study compares the effectiveness and safety of NovoSeven® to FEIBA (FEIBA VH) in haemophilia patients with inhibitors being treated for joint bleeds.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hemophilia A or B with inhibitors to factor VIII or IX, respectively

Max Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2001-09; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Comparison with FEIBA on review of pain, joint mobility and circumference | after 1, 3, 6, and 9 hours of treatment, respectively

SECONDARY OUTCOMES:
Safety variables

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (19):
- United States (19):
  - Novo Nordisk Investigational Site, Little Rock, Arkansas
  - Novo Nordisk Investigational Site, Berkeley, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, New Brunswick, New Jersey
  - Novo Nordisk Investigational Site, Newark, New Jersey
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Hershey, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Houston, Texas

REFERENCES:
- [Result] Young G, Shafer FE, Rojas P, Seremetis S. Single 270 microg kg(-1)-dose rFVIIa vs. standard 90 microg kg(-1)-dose rFVIIa and APCC for home treatment of joint bleeds in haemophilia patients with inhibitors: a randomized comparison. Haemophilia. 2008 Mar;14(2):287-94. doi: 10.1111/j.1365-2516.2007.01601.x. Epub 2007 Dec 10. PMID 18081834
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com